CLINICAL TRIAL: NCT05526690
Title: A Randomized, Open-Label, Two-Period, Crossover Study to Evaluate the Effect of CIN-107 on the Pharmacokinetics of the MATE Substrate, Metformin, in Healthy Subjects
Brief Title: Study to Evaluate the Effect of CIN-107 on the Pharmacokinetics of the MATE Substrate, Metformin, in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIN-107-114
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: Immediate-release metformin (Active Comparator): Treatment A: single 1000 mg dose of immediate-release metformin
  Subjects will be randomly assigned to 1 of 2 sequences: AB or BA.
  * Treatment A: a single 1000 mg dose of immediate-release metformin; and
  * Treatment B: a single 1000 mg dose of immediate-release metformin coadministered with a 10 mg dose of CIN-107.
  All study medication will be administered at 8:00 AM (±2 hours). There will be a minimum 10-day washout between administration of study drug in each treatment period.
  Interventions: Drug: Metformin
- Treatment B: Immediate-release metformin coadministered with a CIN-107 (Experimental): Treatment B: a single 1000 mg dose of immediate-release metformin coadministered with a 10 mg dose of CIN-107
  Subjects will be randomly assigned to 1 of 2 sequences: AB or BA.
  * Treatment A: a single 1000 mg dose of immediate-release metformin; and
  * Treatment B: a single 1000 mg dose of immediate-release metformin coadministered with a 10 mg dose of CIN-107.
  All study medication will be administered at 8:00 AM (±2 hours). For Treatment B, the dose of CIN-107 will be administered 2 hours prior to the dose of metformin.
  There will be a minimum 10-day washout between administration of study drug in each treatment period.
  Interventions: Drug: Metformin; Drug: CIN-107

INTERVENTIONS:
Drug: Metformin — 1000 mg dose of immediate-release metformin
Drug: CIN-107 — 10 mg dose of CIN-107
  Arms: Treatment B: Immediate-release metformin coadministered with a CIN-107

SUMMARY:
This is a randomized, open-label, two-period, crossover Phase 1 to assess the impact of CIN-107 on the pharmacokinetics (PK) of metformin and the safety and tolerability of coadministration of CIN-107 and metformin as compared to metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between the ages of 18 and 55 years, inclusive, at Screening;
* Body mass index between 18 and 30 kg/m2, inclusive;
* In good health based on medical/surgical and psychiatric history, physical examination, electrocardiogram (ECG), vital signs (seated and orthostatic), and routine laboratory tests (serum chemistry, hematology, and urinalysis);
* Normal renal function, defined as estimated glomerular filtration rate ≥85 mL/min/1.73 m2 at Screening and Day -1;
* Nonsmokers who have not used nicotine-containing products (ie, cigarettes, nicotine patch, nicotine chewing gum, or electronic cigarettes) for at least 6 months prior to Screening;

Exclusion Criteria:

* Actively participating in an experimental therapy study; received experimental therapy with a small molecule other than CIN-107 within 30 days of the first dose of study drug or 5 half-lives, whichever is longer; or received experimental therapy with a large molecule within 90 days of the first dose of study drug or 5 half-lives, whichever is longer;
* A personal or family history of long QT syndrome, Torsades de Pointes, other complex ventricular arrhythmias, or family history of sudden death;
* History of, or current, clinically significant arrhythmias, as judged by the Investigator, including ventricular tachycardia, ventricular fibrillation, atrial fibrillation, sinus node dysfunction, or clinically significant heart block. Subjects with minor forms of ectopy (eg, premature atrial contractions) are not necessarily excluded and may be discussed with the Medical Monitor for inclusion;
* Prolonged QT interval corrected by Fridericia's formula (>450 msec);
* Seated systolic blood pressure (BP) >140 mmHg and/or diastolic BP >90 mmHg or systolic BP <90 mmHg and/or diastolic BP <50 mmHg;
* Postural tachycardia (ie, >30 bpm upon standing) or orthostatic hypotension (ie, a fall in systolic BP ≥20 mmHg or diastolic BP ≥10 mmHg upon standing);
* Serum potassium >upper limit of normal (ULN) of the reference range and serum sodium <lower limit of normal of the reference range;
* Aspartate aminotransferase, alanine aminotransferase, or total bilirubin values >1.2 × ULN;
* Positive for human immunodeficiency virus antibody, hepatitis C virus antibody, hepatitis B surface antigen, or severe acute respiratory syndrome coronavirus 2 RNA;
* Evidence or history of any clinically significant immunologic, hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, musculoskeletal, hepatic, psychiatric, neurologic, or allergic (including clinically significant or multiple drug allergies) disease; surgical conditions; cancer (with the exception of basal or squamous cell carcinoma of the skin and cancer that has resolved or has been in remission for >5 years prior to Screening); or any condition that, in the Investigator's opinion, may confound study procedures or results, impact subject safety, or interfere with the absorption, distribution, metabolism, or excretion of the study drug (appendectomy allowed, cholecystectomy prohibited);
* Typical consumption of ≥14 alcoholic drinks weekly; Note: 1 drink of alcohol is equivalent to ½ pint of beer (285 mL), 1 glass of spirits (25 mL), or 1 glass of wine (125 mL).
* Surgical procedures within 4 weeks prior to Check-In (other than minor cosmetic surgery or minor dental procedures) or planned elective surgery during the treatment period;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Up to day 3
  This plasma PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites.
Time to Cmax (Tmax) | Up to day 3
  This plasma PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites.
Area under the concentration-time curve (AUC) from time 0 to 72 hours | Up to day 3
  This plasma PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites.
Maximum plasma concentration (Cmax) of metformin | Up to day 3
  This plasma PK parameter will be determined for metformin.
Time to Cmax (Tmax) of metformin | Up to day 3
  This plasma PK parameter will be determined for metformin.
AUC from time 0 to the time of last quantifiable plasma concentration of metformin | Up to day 3
  This plasma PK parameter will be determined for metformin.
AUC from time 0 to infinity of metformin | Up to day 3
  This plasma PK parameter will be determined for metformin.
Percent of AUC extrapolated of metformin | Up to day 3
  This plasma PK parameter will be determined for metformin.
Terminal phase elimination half-life of metformin | Up to day 3
  This plasma PK parameter will be determined for metformin.
Cumulative amount of metformin excreted in the urine (Ae) of metformin | Up to day 3
  This urine PK parameter will be determined for metformin.
Renal clearance (calculated as Ae/AUC) of metformin | Up to day 3
  This urine PK parameter will be determined for metformin.
Fraction of the dose excreted renally of metformin | Up to day 3
  This urine PK parameter will be determined for metformin.

CONTACTS AND LOCATIONS:
Overall Officials: Leela Leela Vrishabhendra, MD, MD, Principal Investigator — Medpace Clinical Pharmacology Unit
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Background] Freeman MW, Bond M, Murphy B, Hui J, Isaacsohn J. Results From a Randomized, Open-Label, Crossover Study Evaluating the Effect of the Aldosterone Synthase Inhibitor Baxdrostat on the Pharmacokinetics of Metformin in Healthy Human Subjects. Am J Cardiovasc Drugs. 2023 May;23(3):277-286. doi: 10.1007/s40256-023-00572-x. Epub 2023 Feb 15. PMID 36790596
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CIN-107-114&attachmentIdentifier=67f679ad-59a7-42a5-b6e7-ddd9fb0d6985&fileName=CIN-107-114_CSR_synopsis_Redacted.pdf&versionIdentifier=